CLINICAL TRIAL: NCT00563589
Title: A Randomized Single-center Trial of Mycophenolate Mofetil for the Prophylaxis of Graft-versus-host Disease in High Risk Allogeneic Stem Cell Transplantation
Brief Title: Mycophenolate Mofetil for the Prophylaxis of Graft-versus-host Disease in High Risk Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 03-09 R/353; HARECCTR0500036
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Graft vs Host Disease; Hematopoietic Stem Cell Transplantation
Keywords: Acute graft-versus-host disease post high risk allogeneic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Mycophenolic Acid; Methotrexate; Cyclosporine

INTERVENTIONS:
Drug: mycophenolate mofetil, methotrexate, cyclosporin
Drug: Methotrexate and cyclosporin

SUMMARY:
There is a significant (50-80%) risk of acute graft-versus-host disease(GVHD) and early mortality (30%) associated with high risk stem cell transplantation (SCT) such as that from a matched unrelated donor or HLA-mismatch sibling. Mycophenolate mofetil (MMF) has been shown to be an effective and safe immunosuppressant in the prevention and treatment of rejection after solid organ transplantation. Its role in acute GVHD prophylaxis in high risk SCT will be investigated in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing allogeneic SCT with high risk of acute GVHD, ie. from matched unrelated donor or one HLA-locus mismatch sibling

Exclusion Criteria:

* known allergy to mycophenolate mofetil

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-08; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
acute GVHD incidence and grading | 100 Days
chronic GVHD incidence | 3 Years

SECONDARY OUTCOMES:
Mortality, GVHD-related and all cause | 3 Years
Symptomatic side effects attributed to MMF | 60 Days
Date of engraftment | Date of engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence SY Ma, Dr, Principal Investigator — Department of Medicine/ Haematology and Oncology, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, China